CLINICAL TRIAL: NCT05964595
Title: Temporal Diffusion Spectroscopy MRI in Predicting the Comprehensive Positive Score of PD-L1 Expression and the Efficacy of Neoadjuvant Therapy in Head and Neck Squamous Cell Carcinoma
Brief Title: Temporal Diffusion Spectroscopy MRI in Predicting the CPS of PD-L1 Expression and the Efficacy of Neoadjuvant Therapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSKY-2023-498-01
Record Dates: First submitted 2023-06-21; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Magnetic Resonance Imaging; Neoadjuvant Therapy
Keywords: Head and neck squamous cell Carcinoma; Temporal diffusion spectroscopy imaging; Programmed death-ligand 1; Neoadjuvant therapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to explore the application of temporal diffusion spectroscopy MRI in head and neck squamous cell carcinoma (HNSCC).

The main questions it aims to answer are:

* If the quantitative parameters of temporal diffusion spectroscopy MRI can predict the comprehensive positive score (CPS) of pathological PD-L1 expression in HNSCC?
* If the quantitative parameters of temporal diffusion spectroscopy MRI can predict the efficacy of neoadjuvant therapy in HNSCC? Participants will receive head and neck MRI, including T2WI, T1WI, diffusion-weighted imaging (DWI), oscillating gradient spin echo (OGSE) and pulsed gradient spin echo (PGSE) sequence before and after neoadjuvant therapy.

There is not a comparison group in our study.

ELIGIBILITY:
Inclusion Criteria:

* Patients first diagnosed with head and neck squamous cell carcinoma (HNSCC) by pathological biopsy
* Patients proposed to receive 2-3 courses of neoadjuvant chemotherapy and immunotherapy
* Patients without contraindications for MRI, such as nonremovable ferromagnetic metal foreign body, claustrophobia, renal insufficiency, and previous history of gadolinium contrast allergy

Exclusion Criteria:

* Less than 10mm in the maximum diameter of the baseline primary tumor
* Poor MRI image quality with obvious metal or motion artifacts
* The failure to complete the course of neoadjuvant therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients first diagnosed with HNSCC by pathological biopsy and proposed to receive preoperative neoadjuvant therapy at Sun Yat-sen Memorial Hospital
Sampling Method: Non-Probability Sample
Enrollment: 136 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Comprehensive positive score | 1 week before neoadjuvant therapy
  Comprehensive positive score for PD-L1 expression
Pathological response | 1 month after the last neoadjuvant therapy
  Postoperative pathological tumor residual status
Change from maximum transverse tumor diameter after neoadjuvant therapy | 1 week before the first neoadjuvant therapy and 1 month after the last neoadjuvant therapy
  Maximum transverse tumor diameter before and after neoadjuvant therapy

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No